CLINICAL TRIAL: NCT02981160
Title: Validation of a Personal Breath Analyzer for Diet and Energy Expenditure Assessment and Management
Acronym: Breezing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending Organization approval
Sponsor: Banner Health (Other)
Collaborators: Arizona State University (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Flavia Soto, Bariatric Surgeon, Banner Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Breezing Study
Record Dates: First submitted 2016-11-10; First posted 2016-12-05 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care Group (No Intervention): The participants assigned to this group will follow a standard weight loss program for 12-months. This patients will be instructed by the Weight loss program registered dietitian/diet tech in clinic in terms of nutrition regimen, daily intake and calories.Patients will be followed up monthly as per clinic protocol. All visits will include physical measurements including body mass index (BMI) based on height and weight, blood pressure, and body composition (fat percentage). Body composition will be assessed during clinic visits by bio-impedance. Waist circumference (cm) will be measured at the umbilicus.
- Mobile Device Assistant Group (Experimental): This group will follow the same weight loss protocol, monitoring, and clinic visits as the standard weight loss group described above, but will also use the mobile health tool (Breezing) to track REE every visit. This data will be loaded onto an accompanying electronic pad using the Breezing "app" and will be transmitted electronically to the study investigators who will use the information to adjust dietary and physical activity recommendations and targets. The test will be performed at initial visit, 2 weeks, 1, 3, 6 and 12 months after started.
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — The REE testing will be done with the Breezing device, a breath analyzer developed at Arizona State University. The Breezing device is an indirect calorimetry analyzer that measures the rate of oxygen consumption and carbon dioxide production, and determines how much energy the body is burning (REE), and the type of nutrients the body uses to produce energy (energy source). The Breezing device is a cellphone-size, battery-operated, portable technology that syncs with smartphones and electronic pads. The patients will be asked to breathe into a mouthpiece connected to the Breezing device; the data will be then beamed wirelessly to the device. The breath analysis data will displayed on the screen in conjunction with an estimate of total calories burned each day (total energy expenditure, TEE).
  Arms: Mobile Device Assistant Group

SUMMARY:
The purpose of the research is to determine energy expenditure rates and diet and/ physical activity metabolic features of an individual using current state technologies and a new technology created at the Center for Bioelectronics and Biosensors at ASU. This is a pilot study which intent is to validate this device for use in the weight loss patient population.

This study will involve research of metabolic physiological parameters that are measured through the breath of the individuals, together with other physical parameters (weight, height, date of birth, fat and lean body composition via bio-impedance, heart rate, blood pressure, and breathing rate) assessed in the clinic, and a questionnaire about diary physical activities. The study will involve withdrawn of breath samples at resting conditions, and under diets or physical activities regimes.

This instrument will assist our patients in terms of tailoring their diet/nutrition through their weight loss journey prior and after surgery. As a new technology, it will be an excellent tool for compliance assessment and engagement with the Weight Loss Program as well as for long term follow up.

DETAILED DESCRIPTION:
The Breezing® device is a new technology locally invented in the state of Arizona that uses a sensor cartridge and a flow meter to determine the rate of consumed oxygen and produced carbon dioxide in the breath. The sensing technology of the new indirect calorimeter, which used a cell-phone camera as the optical detector. The current Breezing® device uses a code to carry calibration parameters of a single-use sensor cartridge, which can be scanned and recognized by the mobile application (app). The device is 6.0 oz. (170 g), and 1.8 in × 2.1 in × 4.8 in (4.7 cm × 5.4 cm × 12.3 cm), and connects wirelessly to an iOS mobile device, using Bluetooth 4.0 technology.

The mobile device (phone or tablet) receives data from the device, processes information, and then provides test results and summaries through a graphic user interface. It determines the energy expenditure from the measurement of VO2 and VCO2 according to the Weir equation, along with RQ. In addition to the sensor cartridge, the Breezing® device is used with a non-rebreathing 2-valvesmouthpiece.

This new device will provide a more precise information regarding metabolic rate in our Bariatric Patients to better tailor their preoperative diet and monitor their weight loss.

Up to date, this device was never used or validated before in the Bariatric population under this setting.

ELIGIBILITY:
Inclusion Criteria:

* Females or Males between 18 and 50 yo
* Class II and Class III Obesity (BMI 35 and above)

Exclusion Criteria:

- No Obesity. Patients with normal BMI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Improve weight loss measures | 12 months
  Improve weight loss from a standard weight loss program from a mobile breath analyzer device. The device may provide more precise information regarding the metabolic rate in bariatric patients, this device may better tailor patients preoperative diet and assist in monitoring their weight loss.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner Estrella Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: Yes
Baseline and demographic characteristics will be summarized by standard descriptive summaries (e.g. means and standard deviations for continuous variables such as age and percentages for categorical variables such as gender). We will measure differences in weight loss in the two groups using the Mann-Whitney U test